CLINICAL TRIAL: NCT07243522
Title: The Effect of Birth Positions on Pelvic Floor Muscle Strength, Severity, and Quality of Perineal Pain in Primiparous Pregnant Women: A Randomized Controlled Trial
Brief Title: The Effect of Birth Positions on Labor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Emine Demir, Research Assistant (Principal Investigator), Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 25-AKD-139
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Primipara Pregnant; Primipara Labour
Keywords: birth positions; pelvic floor; perineal pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Lithotomy Position Group) (No Intervention)
- Intervention Group (Semi-sitting Position Group) (Experimental)
  Interventions: Other: Semi-sitting birth position

INTERVENTIONS:
Other: Semi-sitting birth position — Pregnant women who present to the maternity unit, meet the inclusion criteria, are assigned to the intervention group after randomization, and agree to participate in the study will be informed about birthing positions by the primary investigator. During the pilot study for the study, it was determined that the ideal position, considering clinical conditions, patient safety, and comfort, is Semi-sittin. Therefore, pregnant women in the intervention group will deliver in the Semi-sitting position.
  Arms: Intervention Group (Semi-sitting Position Group)

SUMMARY:
This study is a randomized controlled trial aimed at evaluating the effects of positions used during labor on pelvic floor muscle strength and the severity and nature of perineal pain in primiparous pregnant women. The World Health Organization (WHO) recommends supporting women's freedom of movement during the second stage of labor and encouraging upright birthing positions. However, in many countries, births are still performed in supine or lithotomy positions, and knowledge and practice regarding upright positions persist. This situation points to a significant knowledge and practice gap for both birthing women and healthcare professionals.

The study will be conducted at the Birth Unit of Bakırçay University Çiğli Training and Research Hospital, Izmir. Following ethics committee approval, the study will be conducted within one year. The sample will consist of 70 primiparous pregnant women who present to the birth unit and meet the inclusion criteria. Participants will be randomly assigned to the intervention and control groups via random.org. Pregnant women in the intervention group will deliver in the Semi-Fowler's (semi-sitting) position, while those in the control group will deliver in the lithotomy position, which is the hospital's standard practice.

Data will be collected in two stages. In the first stage, data will be collected at the onset of labor and when cervical dilation reaches 8-10 cm. In the second stage, data will be collected within 24 hours after delivery, at 6 weeks and 6 months postpartum. Data collection tools will be administered to each woman a total of five times in the first and second stages. Pelvic floor muscle strength will be assessed both objectively with a perineometer and subjectively with the Oxford scale. The severity and nature of perineal pain will be measured with the McGill Pain Scale Short Form.

The hypotheses of the study are that delivering in a semi-sitting position will increase pelvic floor muscle strength and reduce perineal pain. The data will be analyzed using the SPSS 23 software package, using parametric and non-parametric tests. Intention-to-treat (ITT) analysis will be applied when necessary to mitigate the impact of data loss.

This study aims to evaluate not only the effects of birthing positions on the labor process but also their impact on women's health in the postpartum period. This research, which will contribute to expanding the limited literature on this topic, is also expected to support the widespread adoption of a woman-centered approach to care in maternity services.

DETAILED DESCRIPTION:
This study is a randomized controlled trial aimed at evaluating the effects of positions used during labor on pelvic floor muscle strength and the severity and nature of perineal pain in primiparous pregnant women. The World Health Organization (WHO) recommends supporting women's freedom of movement during the second stage of labor and encouraging upright birthing positions. However, in many countries, births are still performed in supine or lithotomy positions, and knowledge and practice regarding upright positions persist. This situation points to a significant knowledge and practice gap for both birthing women and healthcare professionals.

The study will be conducted at the Birth Unit of Bakırçay University Çiğli Training and Research Hospital, Izmir. Following ethics committee approval, the study will be conducted within one year. The sample will consist of 70 primiparous pregnant women who present to the birth unit and meet the inclusion criteria. Participants will be randomly assigned to the intervention and control groups via random.org. Pregnant women in the intervention group will deliver in the Semi-Fowler's (semi-sitting) position, while those in the control group will deliver in the lithotomy position, which is the hospital's standard practice.

Data will be collected in two stages. In the first stage, data will be collected at the onset of labor and when cervical dilation reaches 8-10 cm. In the second stage, data will be collected within 24 hours after delivery, at 6 weeks and 6 months postpartum. Data collection tools will be administered to each woman a total of five times in the first and second stages. Pelvic floor muscle strength will be assessed both objectively with a perineometer and subjectively with the Oxford scale. The severity and nature of perineal pain will be measured with the McGill Pain Scale Short Form.

The hypotheses of the study are that delivering in a semi-sitting position will increase pelvic floor muscle strength and reduce perineal pain. The data will be analyzed using the SPSS 23 software package, using parametric and non-parametric tests. Intention-to-treat (ITT) analysis will be applied when necessary to mitigate the impact of data loss.

This study aims to evaluate not only the effects of birthing positions on the labor process but also their impact on women's health in the postpartum period. This research, which will contribute to expanding the limited literature on this topic, is also expected to support the widespread adoption of a woman-centered approach to care in maternity services.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 35 years of age
* Being primiparous
* Being at term (37-42 weeks)
* Being in the latent phase of the first stage of labor
* Being in the vertex position, having a single, live fetus
* Having an estimated fetal weight between 2500 and 4000 grams
* Having a maternal Body Mass Index <30
* Pregnant women who are expected to give birth vaginally
* Ability to understand and speak Turkish
* Volunteer to participate in the study

Exclusion Criteria:

* Non-cephalic presentation
* Chronic diseases (heart disease, epilepsy, hypertension, hypothyroidism, diabetes, and kidney disease, etc.)
* Risk of obstetric complications (gestational hypertension, cephalopelvic disproportion, antepartum hemorrhage, intrauterine growth restriction, premature rupture of membranes, etc.)
* History of pelvic surgery
* History of prolapse surgery
* History of collagen disorder
* Severe anemia
* Presence of genital tract infection
* Abnormalities of the vulva (presence of vulvar edema, scarring, etc.)
* Application of fundal pressure
* Interventional delivery (use of forceps/vacuum during the second stage, etc.)
* Cesarean section
* Fetal (risk/presence of congenital malformations, estimated fetal weight <2500 g or >4000 g)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-10-07 (Estimated)

PRIMARY OUTCOMES:
Pelvic Floor Muscle Strength Measurement | From enrollment to the end of postpartum at 6 months
  Pelvic floor muscle strength will be assessed both objectively with a perineometer and subjectively with the Oxford scale.

SECONDARY OUTCOMES:
Perineal Pain | From enrollment to the end of postpartum at 6 months
  The severity and nature of perineal pain will be measured with the McGill Pain Scale Short Form.

OTHER OUTCOMES:
Maternal and newborn births outcomes | From enrollment to the end of postpartum at 6 months
  Maternal outcomes such as the duration of the second stage of labor, perineal laceration, and amount of bleeding, and neonatal outcomes such as APGAR score and birth weight will be recorded using the data collection form.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Bakircay University Cigli Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bozkurt M, Yumru AE, Sahin L. Pelvic floor dysfunction, and effects of pregnancy and mode of delivery on pelvic floor. Taiwan J Obstet Gynecol. 2014 Dec;53(4):452-8. doi: 10.1016/j.tjog.2014.08.001. PMID 25510682
- [Result] Catanzarite T, Bremner S, Barlow CL, Bou-Malham L, O'Connor S, Alperin M. Pelvic muscles' mechanical response to strains in the absence and presence of pregnancy-induced adaptations in a rat model. Am J Obstet Gynecol. 2018 May;218(5):512.e1-512.e9. doi: 10.1016/j.ajog.2018.02.001. Epub 2018 Feb 9. PMID 29432755
- [Result] Alperin M, Lawley DM, Esparza MC, Lieber RL. Pregnancy-induced adaptations in the intrinsic structure of rat pelvic floor muscles. Am J Obstet Gynecol. 2015 Aug;213(2):191.e1-7. doi: 10.1016/j.ajog.2015.05.012. Epub 2015 May 13. PMID 25979618
- [Result] Hofmeyr GJ, Vogel JP, Singata M, Habib NA, Landoulsi S, Gulmezoglu AM. Does gentle assisted pushing or giving birth in the upright position reduce the duration of the second stage of labour? A three-arm, open-label, randomised controlled trial in South Africa. BMJ Glob Health. 2018 Jun 29;3(3):e000906. doi: 10.1136/bmjgh-2018-000906. eCollection 2018. PMID 29989055
- [Result] Dabral, A., Pawar, P., Bharti, R., Kumari, A., Batra, A., ve Arora, R. (2018). Upright kneeling position during second stage of labor: a pilot study. Int J Reprod Contracept Obst Gynecol, 7(2), (s.401-407).
- [Result] Berta M, Lindgren H, Christensson K, Mekonnen S, Adefris M. Effect of maternal birth positions on duration of second stage of labor: systematic review and meta-analysis. BMC Pregnancy Childbirth. 2019 Dec 4;19(1):466. doi: 10.1186/s12884-019-2620-0. PMID 31801479
- [Result] Deliktas A, Kukulu K. A meta-analysis of the effect on maternal health of upright positions during the second stage of labour, without routine epidural analgesia. J Adv Nurs. 2018 Feb;74(2):263-278. doi: 10.1111/jan.13447. Epub 2017 Oct 4. PMID 28881046
- [Result] Gupta JK, Sood A, Hofmeyr GJ, Vogel JP. Position in the second stage of labour for women without epidural anaesthesia. Cochrane Database Syst Rev. 2017 May 25;5(5):CD002006. doi: 10.1002/14651858.CD002006.pub4. PMID 28539008
- [Result] Walker KF, Kibuka M, Thornton JG, Jones NW. Maternal position in the second stage of labour for women with epidural anaesthesia. Cochrane Database Syst Rev. 2018 Nov 9;11(11):CD008070. doi: 10.1002/14651858.CD008070.pub4. PMID 30411804
- [Result] Zang Y, Lu H, Zhang H, Zhang X, Yang M, Huang J. Chinese midwives' perceptions on upright positions during the second stage of labour: A qualitative study. Midwifery. 2021 Jul;98:102993. doi: 10.1016/j.midw.2021.102993. Epub 2021 Mar 19. PMID 33823359
- [Result] Zang Y, Lu H, Zhang H, Huang J, Zhao Y, Ren L. Benefits and risks of upright positions during the second stage of labour: An overview of systematic reviews. Int J Nurs Stud. 2021 Feb;114:103812. doi: 10.1016/j.ijnurstu.2020.103812. Epub 2020 Oct 29. PMID 33217662